CLINICAL TRIAL: NCT01413932
Title: A Two-part Study: Part 1 is a Multiple-dose (7-day), Open-label Evaluation of the Safety, Tolerability, and Pharmacokinetics of HT-2157 in Healthy Subjects. Part 2 is a Randomized, Double-blind, Placebo-controlled, Multiple (21-day) Ascending-dose Evaluation of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HT-2157 in Patients With Major Depressive Disorder
Brief Title: Pharmacokinetics - Pharmacodynamic Study of HT-2157 in Healthy Subjects and in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dart NeuroScience, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HT-2157-107
Record Dates: First submitted 2011-08-04; First posted 2011-08-10 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers (Part 1); Major Depressive Disorder (Part 2)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HT-2157 (Experimental)
  Interventions: Drug: HT-2157
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HT-2157 — QD oral dosing
  Arms: HT-2157
Drug: Placebo — QD oral dosing
  Arms: Placebo

SUMMARY:
This is a two part study. The objective of Part 1 is to evaluate the safety, tolerability, and pharmacokinetics of HT-2157 in healthy normal volunteers

Part 2 is a randomized, double-blind, placebo-controlled, multiple (21-day) ascending-dose evaluation of the safety, tolerability, pharmacokinetics, and pharmacodynamics of HT-2157 in patients with major depressive disorder

DETAILED DESCRIPTION:
This is a two part study. The objective of Part 1 is to evaluate the safety, tolerability, and pharmacokinetics of HT-2157 administered for 7-days in healthy normal volunteers

Part 2 is a randomized, double-blind, placebo-controlled, multiple ascending-dose evaluation of the safety, tolerability, pharmacokinetics of HT-2157 administered for 21-days in patients with major depressive disorder. The primary objective of Part 2 is to assess the CNS penetration of HT-2157 in cerebrospinal fluid. In addition, the potential activity of HT-2157 in this patient population may be assessed using exploratory biologic and pharmacodynamic markers of potential efficacy

ELIGIBILITY:
Main Inclusion Criteria (Part 1)

* No clinically relevant abnormalities
* Age 18 to 55 years, inclusive
* Body Mass Index (BMI) of 18.5 to 32 kg/m2

Main Inclusion Criteria (Part 2)

* No clinically relevant abnormalities
* Age 18 to 55 years, inclusive
* Body Mass Index (BMI) of 18.5 to 32 kg/m2
* Mild-to-Moderate major depressive disorder

Main Exclusion Criteria (Part 1)

- Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs

Main Exclusion Criteria (Part 2)

* Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs
* Current and primary Axis I disorder other than MDD

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2011-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
7-day plasma PK profile of HT-2157 | 7-day
  To assess the multiple dose (7-day) plasma PK profile (including AUC, Cmax, Tmax, T1/2, CL/F, Lambda z, VZ/F) of HT-2157 (and its metabolite) administered in the fed state to healthy male and female subjects
To assess the brain penetration of HT-2157 | 21-days
  To assess the brain penetration (PK [including Cmax, Tmax, AUC if possible] in cerebrospinal fluid [CSF]) of HT-2157 (and its metabolite)
PD profile (CSF and peripheral biomarkers, exploratory biologic and pharmacodynamic markers of potential efficacy) of multiple (21-day) doses of HT-2157 patients with MDD | 21-days
  To assess the PD profile (CSF and peripheral biomarkers, exploratory biologic and pharmacodynamic markers of potential efficacy) of multiple (21-day) doses of HT-2157 administered in the fed state to patients with MDD

SECONDARY OUTCOMES:
Safety and tolerability of multiple (7-day) doses of HT-2157 | 7-days
  To assess the safety and tolerability of multiple (7-day) doses of HT-2157 administered in the fed state to healthy male and female subjects. Change from baseline will be assessed for the following measures: Vital signs, 12-lead ECG, laboratory (hematology, chemistry, urinalysis), physical examinations, and adverse events.
Safety and tolerability of multiple (21-day) ascending-doses of HT 2157 | 21-days
  To assess the safety and tolerability of multiple (21-day) ascending-doses of HT 2157 administered in the fed state to patients with MDD. Change from baseline will be assessed for the following measures: Vital signs, 12-lead ECG, laboratory (hematology, chemistry, urinalysis), physical examinations, and adverse events.
21-day ascending-dose plasma PK profile of HT-2157 | 21-days
  To assess the multiple (21-day) ascending-dose plasma PK profile (including AUC, Cmax, Tmax, T1/2, CL/F, Lambda z, VZ/F, RaCmax, RaAUC) of HT-2157 (and its metabolite) administered in the fed state to patients with MDD

CONTACTS AND LOCATIONS:
Overall Officials: Philip Perera, MD, Study Director — Dart NeuroScience, LLC
Locations (1):
- Clinical Site, Glendale, California, United States